CLINICAL TRIAL: NCT00205868
Title: Effectiveness of the Precision Spinal Cord Stimulation System in Patients With Failed Back Surgery Syndrome and Axial Low Back Pain
Brief Title: Spinal Cord Stimulation for Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Lyn Pimentel, Clinical Project Manager, Boston Scientific Corporation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM -SCS -120904
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain
Keywords: Back Pain; Low Back Pain; Chronic Pain; Spinal Cord Stimulation
MeSH Terms: conditions — Chronic Pain; Back Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Precision Spinal Cord Stimulation System — Stimulation on throughout study

SUMMARY:
The purpose of this study is to assess the acute and chronic effectiveness of the Advanced Bionics Precision(TM) Spinal Cord Stimulation System in subjects with failed back surgery syndrome and associated low back axial pain.

Subjects will undergo a temporary or permanent trial to assess their candidacy for placement of an implantable pulse generator. Those who demonstrate a significant clinical reduction in pain will be enrolled in the chronic study. Subjects will be followed for 12 months post implantation to assess the long-term effectiveness of the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for spinal cord stimulation as labeled in the FDA approval for the Precision(R) Spinal Cord Stimulator by Advanced Bionics;
2. Age ≥18 years;
3. Have pain of neuropathic origin;
4. Have chronic pain secondary to surgical spine procedure or intractable low back pain with or without leg pain for at least 3 months and not responding to less invasive clinical procedures.

Exclusion Criteria:

1. Enrollment in any research that would conflict with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramsin Benyamin, MD, Principal Investigator — Millenium Pain Center
Locations (30):
- United States (30):
  - Research Center, Cullman, Alabama
  - Research Center, Daphne, Alabama
  - Research Center, Huntsville, Alabama
  - Research Center, Mesa, Arizona
  - Research Center, Los Angeles, California
  - Research Center, Pasadena, California
  - Research Center, San Diego, California
  - Research Center, Westminster, Colorado
  - Research Center, Jacksonville, Florida
  - Research Center, Jupiter, Florida
  - Research Center, Lewiston, Idaho
  - Research Center, Bloomington, Illinois
  - Research Center, Chicago, Illinois
  - Research Center, Oak Brook, Illinois
  - Research Center, Merrillville, Indiana
  - Research Center, Valparaiso, Indiana
  - Research Center, Boston, Massachusetts
  - Research Center, Pittsfield, Massachusetts
  - Research Center, Rochester, Minnesota
  - Research Center, Billings, Montana
  - Research Center, Winston-Salem, North Carolina
  - Research Center, Hamilton, Ohio
  - Research Center, Eugene, Oregon
  - Research Center, Allentown, Pennsylvania
  - Research Center, Philadelphia, Pennsylvania
  - Research Center, Spartanburg, South Carolina
  - Research Center, Murray, Utah
  - Research Center, Provo, Utah
  - Research Center, Cudahy, Wisconsin
  - Research Center, Rice Lake, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Efforts were made but the information is not accessible at this time. Hence assignment not available.
Groups:
- Spinal Cord Stimulation: Subjects will undergo a temporary or permanent trial to assess their candidacy for placement of an implantable pulse generator. Those who demonstrate a significant clinical reduction in pain will be enrolled in the chronic study. Subjects will be followed for 12 months post implantation to assess the long-term effectiveness of the therapy.
Period: Overall Study
Arm/Group | Spinal Cord Stimulation
Started | 304
Completed | 304
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Efforts were made but the information is not accessible at this time. Hence baseline measures not reported.
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of SCS Stimulation in Reducing Back Pain Associated With Failed Back Surgery Syndrome After 12 Months of Use.
Description: Effectiveness of SCS stimulation in reducing back pain associated with Failed Back Surgery Syndrome after 12 months of use as measured by 0 - 10 numerical rating scale (Numerical Rating Scale, NRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine"
Time Frame: 1 year
Population: Efforts were made but the information is not accessible at this time. Hence outcome measures not reported.
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 0

2. Primary Outcome: Effectiveness of SCS Stimulation in Reducing Leg Pain Associated With Failed Back Surgery Syndrome After 12 Months of Use.
Description: Effectiveness of SCS stimulation in reducing leg pain associated with Failed Back Surgery Syndrome after 12 months of use as measured by 0 - 10 numerical rating scale (Numerical Rating Scale, NRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine"
Time Frame: 1 year
Population: Efforts were made but the information is not accessible at this time. Hence outcome measures not reported.
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Patients Who Achieve a Significant Clinical Reduction in Back Pain Defined as >50% Reduction in VAS Score With Stimulation Compared With no Stimulation
Time Frame: 1 year
Population: Efforts were made but the information is not accessible at this time. Hence outcome measures not reported.
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through end of study.
Description: Efforts were made but the information is not accessible at this time. Hence adverse events not reported.
Arm/Group | Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/304
Serious Adverse Events (participants affected / at risk) | 0/304
Other Adverse Events (participants affected / at risk) | 0/304

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes